CLINICAL TRIAL: NCT07129980
Title: Refractive and Visual Outcomes With the ARGOS Biometer In Eyes With a History of Refractive Surgery: ARGOS Study
Status: Completed | Type: Observational
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Other Study IDs: ARGO-IIT
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cataract
Keywords: Biometry, IOL Calculations
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Participants: Eligible participants were subjects with a history of prior myopic corneal refractive surgery as confirmed by preoperative corneal topography and imaging. All subjects included in the study underwent traditional cataract surgery with a 2.4 millimeter (mm) corneal incision and were implanted with a standard monofocal intraocular lens. Following the procedure, subjects returned at 8-12 weeks postoperative for a study visit in which a manifest refraction was performed.
  Interventions: Device: ARGOS Biometer

INTERVENTIONS:
Device: ARGOS Biometer — The ARGOS biometer uses swept-source optical coherence tomography (SS-OCT) with a 1060 nm tunable laser to capture high-resolution B-scan images of the entire eye. This technology enables sum-of-segments (S-O-S) biometry, measuring each ocular component-corneal thickness, aqueous depth, lens thickness, and vitreous length-individually and summing these values to determine total axial length. SS-OCT provides deep tissue penetration while simultaneously capturing keratometry, white-to-white, and pupillometry data in a single scan. For keratometry measurements, the ARGOS uniquely employes SS-OCT-based telecentric keratometry, which involves projection of 16 infrared LEDs in a wider 3.0 mm ring pattern onto the cornea and calculates curvature from those reflections.
  Other Names: Swept Source Optical - Optical coherence tomography (SS-OCT)

SUMMARY:
The study is to evaluate the visual and refractive outcomes in eyes with prior myopic refractive surgery undergoing cataract surgery for intraocular lens (IOL) power calculations.

DETAILED DESCRIPTION:
This was a prospective, single-site, study evaluating the accuracy of the ARGOS biometer in subjects with a history of myopic corneal refractive surgery including Laser-Assisted In Situ Keratomileusis (LASIK) and Photorefractive Keratectomy (PRK).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated cataract surgery with a history of myopic corneal laser refractive surgery
* Subjects electing to undergo implantation with a monofocal/non-toric IOL
* Willing and able to comprehend informed consent and complete an 8-week visit.
* Potential postoperative Corrected Distance Visual Acuity (CDVA) of 20/20 or better in each eye based on Investigator's medical opinion

Exclusion Criteria:

* Concurrent or prior ocular surgery within the previous 12 months.
* Ocular comorbidity that could reduce the potential postoperative CDVA based on the discretion of the operating surgeon
* History of hyperopic laser corneal refractive surgery
* History of radial keratotomy
* Irregular corneal astigmatism or keratoconus 6. Eyes with intraoperative or postoperative complications 7. Eyes with BCDVA worse than 20/100 preoperatively 8. Subjects who are pregnant or plan to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or females undergoing uncomplicated cataract surgery with a history of myopic corneal laser refractive surgery and subjects electing to undergo implantation with a monofocal/non-toric IOL
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Refractive Outcomes | 12 weeks
  To evaluate refractive outcomes in eyes with prior myopic refractive surgery undergoing cataract surgery using Sum-of-Segment biometry for IOL power calculations.
Visual Outcomes | 12 weeks
  To evaluate visual in eyes with prior myopic refractive surgery undergoing cataract surgery using Sum-of-Segment biometry for IOL power calculations.

CONTACTS AND LOCATIONS:
Overall Officials: John Berdahl, MD, Principal Investigator — Vance Thompson Vision Clinic Prof. LLC
Locations (1):
- Vance Thompson Vision Clinic, Prof. LLC, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No